CLINICAL TRIAL: NCT01178164
Title: Prevalence of Fabry's Disease in a Population of Patients With Chronic Pains
Acronym: DOUFAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2010/04
Record Dates: First submitted 2010-08-04; First posted 2010-08-10 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Pain; Fabry's Disease
Keywords: chronic pains; unknown aetiology
MeSH Terms: conditions — Pain; Fabry Disease; Chronic Pain | interventions — Blood Specimen Collection; Biological Products; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnosis of Fabry disease (Experimental)
  Interventions: Genetic: Blood sampling for biological and genetic analysis

INTERVENTIONS:
Genetic: Blood sampling for biological and genetic analysis — * Clinical examination
  * Blood sampling for biochemical enzymatic measures of alphagalactosidase A activity in males, and genetic analysis using direct sequencing of GLA in females.

SUMMARY:
Fabry disease (FD) is a rare X-linked multisytemic lysosomal disorder caused by alpha-galactosidase deficiency. Globotriaosylcéramide (Gb3) deposits are observed in almost all tissues examined. Signs of the disease appear earlier and are more severe in affected males than in females. Myocardiopathy, renal failure and neurological signs including chronic pain and peripheral neuropathies are the most frequent signs. The availability of two enzymatic replacement therapies now provides a specific and effective treatment for patients. The prevalence of FD is estimated between 1/40,000 and 1/117,000. The frequency of Fabry disease has previously been estimated in several series of patients presenting one single sign, ie renal failure, hypertrophic myocardiopathy and early onset stroke. However, no data are available about the prevalence of FD in populations of patients suffering from chronic pains of unknown origin.

The diagnosis of FD will be performed by standard procedures following international recommendations. These require the search for a deficiency of alphagalactosidase A activity on leucocytes in males and genetic analysis of the GLA gene in females (Lidove et al. 2007).

The patients in whom the diagnosis of FD is established during this study, will be call in for an additional visit in the Investigating Centre in order to confirm the diagnosis and propose suitable assessment and care.

ELIGIBILITY:
Inclusion Criteria:

* patients of both sex
* aged from 6 to 65
* with chronic pains of unknown aetiology including:
* acroparesthesias
* and/or pain crises evolving more than 3 months
* continued neuropathic evolving more than 3 months
* and/or multiple pains evolving more than 3 months
* and/or recurrent abdominal crises of pain who come for a clinical visit in the Centre Douleurs Chroniques in the CHU of Bordeaux.

Exclusion Criteria:

* chronic pain of known cause

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Fabry disease in one patient suffering from chronic pains | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Virginie DOUSSET, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Centre Douleurs Chroniques, Hopital Pellegrin, Bordeaux, France